CLINICAL TRIAL: NCT04484129
Title: Multidrug Resistant Tuberculosis Close Contacts Tracing in China
Brief Title: MDR-TB Close Contacts Tracing in China (TCCT Study)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Other Study IDs: KY2020-806
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Multidrug Resistant Tuberculosis
Keywords: Multidrug Resistant Tuberculosis; latent tuberculosis; close contacts; transmission
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Close contacts of MDR-TB patients: Close contacts of MDR-TB who met the inclusion and exclusion criteria were enrolled. Routine follow-up is scheduled at week 8, 20, 32, and 80. During the visit, participants with suspected tuberculosis symptoms will have detailed clincial assessent, weight measurement, sputum smear, sputum culture and drug sensitivity examination, imaging examinations, etc. For patients diagnosed with TB, the trial ends. Proper treatment will be started. For all paricipants who are not diagnosed with tuebrculosis in previous follow-up, the last follow-up of this study is all "face-to-face" visits. Sputum smear, sputum culture and chest imaging screening will be performed when necessary to exclude the possibility of tuberculosis infection. In addition, If the participants has suspected TB symptoms or is diagnosed with TB in another hospital, the researchers can be contacted for follow-up at any time.

SUMMARY:
To investigate the incidence of etiologically confirmed or clinically diagnosed active tuberculosis in close contacts of MDR-TB patients.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study. MDR-TB patients from multi-centers in China were continuously evaluated one by one, their close contacts were screened for elibgility. All subjects were followed for the same length of time: 80 weeks after enrollment. The symptoms and signs of tuberculosis were followed up to monitor the occurrence of tuberculosis.

The primary objective is to investigate the incidence of etiologically confirmed or clinically diagnosed active TUBERCULOSIS in close contacts of MDR-TB patients.

The secondary objective is to assess latent TB infection rates in close contacts of MDR-TB patients; evaluate the high risk factors of TUBERCULOSIS in close contact population; assess the loss rate of close contacts within 80 weeks; assess the 80-week mortality rate among close contacts; isolate the mycobacterium tuberculosis from all patients with active tuberculosis and analyze drug resistance to evaluate the homology and drug-resistant transmission pattern of Mycobacterium tuberculosis.

ELIGIBILITY:
The index patient:

Inclusion Criteria:

1.18-70 years old; 2.Has smear-positive pulmonary tuberculosis with initial laboratory results with resistance to rifampicin confirmed by GeneXpert; 3.Have an identifiable address and stay in the area during the study period.

Exclusion Criteria:

1. Combined extrapulmonary tuberculosis;
2. HIV antibody positive and AIDS patients;
3. Critically ill patients, and according to the judgment of the research physician, it is impossible to survive for more than 4 months.

Termination/termination criteria:

1. The patient requests to withdraw from the visit;
2. Misdiagnosis and error.

The close contacts:

Inclusion Criteria:

1. Willing to participate in trial treatment and follow-up and can give informed consent;
2. Willing to carry out HIV testing;
3. More than 6 hours of cohabitation per week in the 2 weeks prior to diagnosis of the index case.

Exclusion Criteria:

1. Patients with active tuberculosis confirmed clinically or etiologically;
2. Mental illness and severe neurosis;
3. The researchers determined that there were any ineligible conditions.

Termination/termination criteria:

1. The patient requests to withdraw from the visit;
2. Find a violation of inclusion or exclusion criteria during treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population enrolled in this study is close contact of patients with MDR-TB
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-21 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed cases of active tuberculosis | 80 weeks after enter the group
  Mycobacterium tuberculosis was indicated to be positive by etiology, and the positive ones were confirmed by molecular identification. A false positive may be determined if the investigator determines that the etiological diagnosis is inconsistent with the patient's clinical condition, or that the patient's symptoms, signs, or influence of the medical diagnosis has not responded to treatment.
Clinical diagnosis of active tuberculosis | 80 weeks after enter the group
  History, signs, imaging studies (mainly chest CT), or other diagnostic methods suggest objective evidence (cough, fever, night sweats, wasting, hemoptysis) for the diagnosis of tuberculosis, rather than other diseases.

SECONDARY OUTCOMES:
Incidence of latent tuberculosis infection | at enrollment
  Incidence of latent tuberculosis infection at enrollment
Risk factors associated with TB development | 80 weeks after enter the group
  Risk factors associated with TB development among the close contact population
Compliance of follow-up | 80 weeks after enter the group
  number of participants who complete the follow-up schedule
Comparison the Mycobacteria tuberculosis strains between index patients and their contacts | 80 weeks after enter the group
  All Mycobacteria tuberculosis strains from index patients ans close contacts will be analyzed to explore the transmission pattern

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, PhD, Principal Investigator — Huashan Hospital
Locations (8):
- China (8):
  - The Third People's Hospital of Shenzhen City, Shenzhen, Guangzhou
  - Guiyang Public Health Treatment Center, Guizhou, Guizhou
  - Henan Hospital of Infectious Diseases, Zhengzhou, Henan
  - Jiangxi Public Health Center, Nanchang, Jiangxi
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Chest Hospitalof Xinjiang Uygur Autonomous Region of PRC, Ürümqi, Xinjiang
  - Hangzhou Red Cross Hospital, Hangzhou, Zhejiang
  - The Central Hospital of Wenzhou City, Wenzhou, Zhejiang